CLINICAL TRIAL: NCT06569745
Title: Primary School Children's Oral and Dental Health Knowledge Assessed With Different Educational Methods: A Cross-Sectional Study
Brief Title: Evaluation of Children's Oral Health Education With Different Education Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Canan Bayraktar Nahir, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-KAEK-275
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries in Children
Keywords: dental health education; primary school; children; video-audio demonstration; peer influence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verbal Explanation Group (Experimental): Verbal Explanation Group
  Interventions: Other: Verbal Explanation
- Animation Group (Experimental): Animation Group
  Interventions: Other: Animation Video Display
- Peer-Led Reels Group (Experimental): Peer-Led Reels Group
  Interventions: Other: Peer-Led Reels Video Display

INTERVENTIONS:
Other: Verbal Explanation — In the verbal explanation group, a researcher wearing white coat provided oral and dental health education for 3 minutes using a jaw model
  Arms: Verbal Explanation Group
Other: Animation Video Display — In the animation group, oral and dental health education was presented to the children in the form of a cartoon lasting 1 minute and 17seconds. The animation video was created by the researcher using the test version of "www.vyond.com". The animation featured a character voiced by one of the researchers, informative texts, and background music. The character conveyed information about oral and dental health education, using both voice and text content.
  Arms: Animation Group
Other: Peer-Led Reels Video Display — In the peer-led reels group, oral and dental health information was presented for 1 minute using a video created on the Instagram platform. The video showed oral hygiene information being provided to a child of a similar age to the target audience with the child then demonstrating the behaviour with music in the background. The video included some text, but did not feature the child's voice or information.
  Arms: Peer-Led Reels Group

SUMMARY:
Different educational methods may play a crucial role in oral and dental health education programs.

The aim of our study is to evaluate the effects of different educational methods on the knowledge levels of primary school children regarding oral and dental health. The null hypothesis of this study is that there is no difference between education methods on the level of knowledge acquired by children about oral and dental health.

DETAILED DESCRIPTION:
This cross-sectional study included 10-11 year old 5th grade students from primary schools located in the center of Tokat, Turkey. The purpose of the study was explained to the school principal, and after obtaining their approval, informed consent forms were sent to the parents. The study was conducted between January and June 2022 in conference halls or classrooms within the schools.

The study questions were developed by 4 expert pediatric dentists after a thorough literature review. The questions were designed to test the children's knowledge of oral and dental health. The questionnaire was divided into two parts. The first part collected demographic data, such as age, gender, and tablet/mobile phone usage. The second part consisted of 8 questions assessing general knowledge about oral and dental health. Each correct answer was scored as 1 point, while incorrect and unanswered questions received 0 points.

In the verbal explanation group, a researcher wearing white coat provided oral and dental health education for 3 minutes using a jaw model.

In the animation group, oral and dental health education was presented to the children in the form of a cartoon lasting 1 minute and 17seconds. The animation video was created by the researcher using the test version of "www.vyond.com". The animation featured a character voiced by one of the researchers, informative texts, and background music. The character conveyed information about oral and dental health education, using both voice and text content.

In the peer-led reels group, oral and dental health information was presented for 1 minute using a video created on the Instagram platform. The video showed oral hygiene information being provided to a child of a similar age to the target audience with the child then demonstrating the behaviour with music in the background. The video included some text, but did not feature the child's voice or information.

All educational methods included the same information about general oral and dental health. Following the education, the children completed the same questionnaire again.

Statistical Analysis Data analysis was conducted using the IBM Statistical Package for the Social Sciences (SPSS for Windows, version 26.0, SPSS Inc., Chicago, IL, USA). Descriptive statistics including number and percentage for categorical data and mean and standard deviation for continuous data were calculated. The normality of the data was assessed using the Kolmogorov-Smirnov test. The Wilcoxon test was used to compare the knowledge levels before and after dental education, while the analysis of covariance (ANCOVA) was used to evaluate the effects of group, gender, and tablet/mobile phone usage on the knowledge level at the end of the oral and dental health education. A p-value of <0.05 was considered statistically significant in all tests.

ELIGIBILITY:
Inclusion Criteria:

Children aged 10-11 years

Exclusion Criteria:

Mental, visual, or auditory disabilities Not being diagnosed with a syndrome

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
After education knowledge | 1 year
  A questionnaire was administered to the children to measure their oral and dental health knowledge and then educations were given. After the educations, the same questionnaire was applied again to determine how effective these educations were according to the groups and their knowledge levels were evaluated.
  The questionnaire was divided into two parts. The first part collected demographic data, such as age, gender, and tablet/mobile phone usage. The second part consisted of 8 questions assessing general knowledge about oral and dental health. Each correct answer was scored as 1 point, while incorrect and unanswered questions received 0 points.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Bayraktar Nahir, Principal Investigator — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
with the link to be prepared later
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Unlimites
Access Criteria: no criteria

REFERENCES:
- [Derived] Bayraktar Nahir C, Cosgun A, Sahin ND, Altan H. Primary school children's oral hygiene knowledge assessed with different educational methods: a cross-sectional study. BMC Oral Health. 2025 Jan 28;25(1):148. doi: 10.1186/s12903-025-05493-6. PMID 39875880